CLINICAL TRIAL: NCT01324934
Title: Prospective, Randomized, Multi-center, Open Label, Phase III Study to Evaluate the Efficacy and Safety of Immunosuppression Following a Heart-beating Cadaveric Renal Transplantation Based on the Use of Rabbit Anti-T-lymphocyte Serum, Tacrolimus and Mycophenolate, Free of Concomitant Corticosteroids From the Start of Immunosuppression
Brief Title: Efficacy and Safety of ATG-Fresenius Following a Renal Transplantation, Without Corticosteroids
Acronym: IBERICA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment became very slow.
Sponsor: Neovii Biotech (Industry)
Collaborators: Eurotrials Brasil Consultores Cientificos Ltda (Industry); Recerca Clínica S.L. (Industry); PsyConsult (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP-AS-24-ES
Record Dates: First submitted 2011-03-21; First posted 2011-03-29 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Renal Transplant Rejection
Keywords: acute rejection; chronic rejection; subclinical rejection; renal transplantation; steroid-free; kidney transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group (Active Comparator): immunosuppressive treatment consisting of ATG-Fresenius/TAC/MMF or Myfortic
  Interventions: Drug: ATG-Fresenius S
- Control Group (No Intervention): immunosuppressive treatment consisting of TAC, MMF or Myfortic, and corticosteroids.

INTERVENTIONS:
Drug: ATG-Fresenius S — Dosage: Single high-dose of 9 mg/kg pre-operatively, followed by 3 mg/kg/d at day +2 and +4. ATG-Fresenius treatment at Days 0, +2, and +4 is mandatory.
  (In case of persisting DGF, the treatment is left to the discretion of the investigator. Treatment options include the continuation of ATG-Fresenius treatment with 3 mg/kg/d at Day +6 and if deemed necessary also at Day +8 - but without corticosteroids).
  Arms: Study Group

SUMMARY:
The main objective of the study is the assessment of the overall graft rejection rate (acute, chronic and subclinical) between a treatment with ATG-Fresenius administered in addition to standard treatment consisting of CellCept® or Myfortic®/TAC and without corticosteroids and a treatment consisting of CellCept® or Myfortic®/TAC and corticosteroids during the first year after renal transplantation.

ELIGIBILITY:
Inclusion Criteria

* Signed and dated informed consent form,
* End-stage renal disease,
* Candidates for a first transplantation,
* Re-transplant patients are eligible if a graft loss after transplantation was NOT due to immunological reasons,
* Availability of a heart-beating cadaveric donor up to 70 years of age with a cold ischemia time shorter than 36 hours,
* Male or female patients between 18 to 75 years of age inclusive,
* Patients able to comply with all study related requirements,
* Patients able to receive oral medication,
* Women of childbearing age with a safe contraceptive method throughout the study.

Exclusion Criteria

* Women who are pregnant or breast feeding,
* Known Human Immunodeficiency Virus,
* Hepatitis B Virus or Hepatitis C Virus infection,
* Severe actual viral, bacterial or fungal infection not adequately controlled,
* Patients with anamnestically known hypersensitivity to rabbit immunoglobulin antibodies or positive rabbit immunoglobulin skin test or known allergies to any component of the immunosuppressive drugs per protocol,
* Patients at high immunological risk defined as current PRA > 25% or historical PRA > 50%,
* Patients receiving pre-transplant immunosuppressive treatment, including corticosteroids,
* Patients with current or history of malignancies (exception basal cell carcinoma or squamous cell carcinoma in remission),
* Patients with previous transplantation except 1st graft loss due to surgical complications,
* Patients receiving combined transplantation,
* Patients with major organ dysfunctions,
* Serious psychiatric or psychological disorders,
* Pre-transplant thrombocytopenia: < 50,000 thrombocytes/µl, Pre-transplant leukopenia: < 2,000 leukocytes/µl,
* Unable or unwilling to comply fully with the protocol,
* Participation in another study of an investigational medicinal product concurrently or within the last 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the incidence of biopsy-proven acute allograft rejection after 12 months, including all types of rejections like: • acute rejection • chronic rejection • subclinical rejection | 1 year

SECONDARY OUTCOMES:
Time of onset, histological severity and incidence of steroid resistance of acute and chronic rejections | 1 year
Incidence and duration of initial DGF | 1 year
Renal function | 1 year
Patient and Graft survival | 1 year
Safety endpoints are the incidence of AEs/SAEs and ADRs | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Rengel, Dr, Principal Investigator — Hosptial Gregorio Maranon, Madrid, Spain
Locations (10):
- Portugal (4):
  - Centro Hospitalar de Lisboa Ocidental, Carnaxide
  - Hospitais da Universidade de Coimbra, Coimbra
  - Hospital de Curry Cabral, Lisbon
  - Hospital Geral de Santo António, SA, Porto
- Spain (6):
  - Hospital Universitario Juan Canalejo, A Coruña
  - Hospital Universitari Clinic i Provincial, Barcelona
  - Hosptial Gregorio Maranon, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid